CLINICAL TRIAL: NCT03444909
Title: CIPTEx : Collection of Information by Tocography External
Brief Title: Collection of Information by Tocography External
Acronym: CIPTEx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioSerenity (Industry)
Collaborators: Pitié-Salpêtrière Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017-A03123-50
Record Dates: First submitted 2018-01-04; First posted 2018-02-26 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Pregnancy Related
Keywords: Monitoring

STUDY DESIGN:
Intervention Model Description: 35 women will be divided into 3 test groups. results will be analyse in fonction of the repartition of the gestationnal age
  10 women between 24-29 Week of amenorrhea (WA); 15 women between 30-35 WA; 10 women between 36-41 WA will be included.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- cardiotocograph and Toconaute (Experimental): monitoring with cardiotocograph and next with the Toconaute of Bioserenity
  Interventions: Device: cardiotocograph; Device: Toconaute
- Cardiotocograph and Toconaute and Electrophysiological device (Experimental): monitoring withardiotocograph and next with Toconaute and next with the electrophysiological device
  Interventions: Device: cardiotocograph; Device: Toconaute; Device: electrophysiological device (Micromed)
- Cardiotocograph and electrophysiological device (Experimental): monitoring with the cardiotocograph and next with the electrophysiological device (Micromed)
  Interventions: Device: cardiotocograph; Device: electrophysiological device (Micromed)

INTERVENTIONS:
Device: cardiotocograph — Monitoring of 20 min with the cardiotocograph
Device: Toconaute — Monitoring of 20 min withToconaute
  Arms: Cardiotocograph and Toconaute and Electrophysiological device; cardiotocograph and Toconaute
Device: electrophysiological device (Micromed) — Monitoring of 20 min with the cardiotocograph
  Arms: Cardiotocograph and Toconaute and Electrophysiological device; Cardiotocograph and electrophysiological device

SUMMARY:
The purpose of this trial is to create a comparative database, with data obtained with a new monitoring device of pregnant women,Toconaute, and two standard : a clinical cardiotocograph,and an electrophysiological signal medical device. It will allow to optimize the development of this new device.

The use of the Toconaute and/or the electrophysiological medical device will succeed to the usual monitoring of pregnant women with a cardiotocograph. It will not change their medical care.

The trial will include up to 35 pregnant women between 24 and 41 weeks of amenorrhea that requires discontinuous monitoring. It will last about 12 months, with an estimated inclusion period of 11 month.

DETAILED DESCRIPTION:
The main objective is to compare measurements for different gestational age, between: the standard cardiotocograph with those of our device, or between the standard cardiotocograph and the Toconaute and the electrophysiological device, or between the Toconaute and the electrophysiological device.

As a second objective, we want to build a database between the cardiotocograph, the Toconaute and the electrophysiological device, to optimize the development of the Toconaute device.

The trial will include up to 35 healthy adult women pregnant between 24 and 41 weeks of amenorrhea requiring discontinuous monitoring. The trial will not change the usual medical management of women, the Toconaute device will be tested following their usual monitoring. The trial will last approximately 12 months, with an estimated inclusion period of 11 months.

In order to be able to identify possible adverse effects related to the device, women participating simultaneously in another clinical trial can not be included. A delay of 1 month minimum after participation in another clinical trial is requested.

The risks associated with the use of the Toconaute in the trial are considered low and acceptable.

Participating women will receive information from the investigator or the midwife who represents it, and will cover all the points provided for in Article L1122-1. They will be informed of the risks and their right to refuse to participate in a search or to withdraw their consent at any time without incurring any liability or prejudice. Women wishing to participate will receive the newsletter and then sign a consent. A copy of the consent will be issued to them.

As part of the test, the care of the pregnant woman is not changed, the use of the Toconaute will succeed to their usual monitoring with a cardiotocograph. The investigating physician or midwife will therefore follow the recommendations of the usual medical procedure regarding measurements performed by external cardiotocography.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women adult (> 18 years) from 24 to 41 weeks of amenorrhea with or without contractions
* Requiring an intermittent monitoring (including women parturient in pre-labour)
* speaking and understanding well French
* Affiliated to a social security system

Exclusion Criteria:

* Multiple pregnancy
* Women requiring a continuous monitoring (in advanced labour)
* Refusal of consent
* Minors
* Wounds on the stomach
* Women under protection or person not capable of following the procedure of use (according to the judgment of the investigator)
* Allergy known about the silver, the polyamide, the synthetic materials, a component of STIMEX gel.
* Use of device on people who the compression of a garment tightened on the stomach could cause pains, respiratory problems or worsening of the health
* Person equipped with a device of electric stimulation;
* Current participation in a clinical trial or participation in a previous clinical trial including a period of not past deficiency of 1 month at the time of this clinical trial.
* Use of the device within for a resuscitation or intensive care
* person with a defibrillator, a stimulating one of the vagus nerve, or high-frequency surgical device.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-12-11 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-12-11 (Actual)

PRIMARY OUTCOMES:
comparison of measures from Toconaute, cardiotocograph and Micromed device | 1 year
  evaluation of the quality of signal (heart rate of mother and foetus, electrocardiogramme mother and foetus, contractions)

SECONDARY OUTCOMES:
creation of a comparative database between the cardiotocograph and the toconaute and the electrophysiological device (micromed) | 1 year
  databases will be created comparing data from cardiotocograph and data from toconaute and data from the electrophysiological device

CONTACTS AND LOCATIONS:
Locations (1):
- Salpêtrière Hospital, Paris, France